CLINICAL TRIAL: NCT05184413
Title: Effectiveness of a Multimodal Telerehabilitation Program Combining Pain Neuroscience Education and Therapeutic Exercise for Patients With Carpal Tunnel Syndrome: A Randomized Controlled Trial
Brief Title: Telerehabilitation in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clínico La Florida (Other)
Collaborators: University of Chile (Other); University of Valencia (Other); Hospital San José (Unknown); Hospital Provincia Cordillera (Unknown)
Responsible Party: Principal Investigator, Rodrigo Ignacio Nunez Cortes, Principal Investigator, Hospital Clínico La Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RNCHLF0022020
Record Dates: First submitted 2021-11-27; First posted 2022-01-11 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: pain; disability; education; exercise
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain; Motor Activity | interventions — Combined Modality Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator at each center responsible for conducting the study evaluations will be blinded to group assignment. A second investigator will be responsible for generating randomization, sequencing, enrolling participants, and assigning participants to treatment. Patients will be blinded to the assigned group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal treatment (Experimental): Therapeutic Exercise plus Pain Neuroscience Education
  Interventions: Other: Multimodal treatment
- Unimodal treatment (Active Comparator): Therapeutic Exercise
  Interventions: Other: Unimodal treatment

INTERVENTIONS:
Other: Multimodal treatment — A multimodal telerehabilitation intervention will be conducted through Whatsapp video calls. The combined treatment includes: 1) One 30-minute session of education in neurosciences of pain, using audiovisual material with examples and metaphors to improve the patient's understanding. In addition, two sessions of reinforcement of key contents will be held every 15 days; 2) Therapeutic exercise program: active wrist and finger exercises, stretching, mobilization exercises of the median nerve, and aerobic exercise (brisk walking). Each exercise will be dosed on a personalized basis, with a perceived exertion of 4-5 on the Borg scale. Therapeutic exercise will be self-administered, 3 sessions per week for 6 weeks. Telerehabilitation sessions will be performed every 15 days to monitor adherence and adjust the exercise dose.
  Arms: Multimodal treatment
Other: Unimodal treatment — An unimodal telerehabilitation intervention will be performed through Whatsapp video calls. The treatment will include only a therapeutic exercise program: active wrist and finger exercises, stretching, mobilization exercises of the median nerve, and aerobic exercise (brisk walking). Each exercise will be dosed on a personalized basis, with a perceived exertion of 4-5 on the Borg scale. Therapeutic exercise will be self-administered, 3 sessions per week for 6 weeks. Telerehabilitation sessions will be performed every 15 days to monitor adherence and adjust the exercise dose.
  Arms: Unimodal treatment

SUMMARY:
Carpal tunnel syndrome (CTS) is a compressive peripheral neuropathy characterized by pain, tingling sensation and paresthesia in the territory of the median nerve. These symptoms cause significant functional impairment that affects patients' quality of life. Pain neuroscience education (PNE) combined with therapeutic exercise (TE) has shown good results in patients with chronic pain, but the effects of this multimodal treatment via telerehabilitation have not been studied in patients with CTS. Telerehabilitation has demonstrated clinical and functional outcomes as effective as face-to-face interventions, being a good alternative to improve accessibility to rehabilitation care in a context of pandemic and social distancing. The purpose of this study is to provide coordinated, patient-centered care by implementing a Telerehabilitation model for patients with severe CTS. The objective of this study was to compare the effectiveness of a multimodal therapy program (TE plus PNE) versus a unimodal treatment (TE) in patients with CTS.

A Randomized Controlled Trial, simple-blind and multicenter study will be conducted. Patients will be randomly assigned to the multimodal treatment group (TE plus PNE) or to the unimodal treatment group (TE). At admission, an investigator blinded to treatment assignment will conduct data collection. The measurements will be the following outcomes: a) Pain Catastrophizing Scale; b) Tampa Scale for Kinesiophobia-11; c) Numerical Rating Scale (NRS); d) Boston Carpal Tunnel Questionnaire; e) Hospital Anxiety and Depression Scale; f) Quality of Life, using the EQ-5D instrument; g) Patient's global impression of change; h) Katz Diagram; These evaluations will be performed again at week 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years of age, severe CTS medical diagnosis, duration of symptoms for more than three months, access to a smartphone with internet, and acceptance to participate in the study.

Exclusion Criteria:

* Inability to understand instructions, non-controlled mental health pathology, cognitive problems and previous surgery in the upper limb.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain Catastrophizing Scale (PCS) at 6 and 12 weeks | Baseline (0 weeks), 6 weeks and 12 week
  To assess catastrophic thinking as a response to pain through 13 statements with 4 possible options from 1 "not at all" to 4 "all the time". a higher score indicates a higher catastrophic thinking
Change from Baseline Tampa Scale for Kinesiophobia-11 (TSK-11) at 6 and 12 weeks | Baseline (0 weeks), 6 weeks and 12 week
  Kinesiophobia will be evaluated by Tampa Scale for Kinesiophobia (TSK-11SV) (Spanish adaptation. Gómez-Pérez, López-Martínez y Ruiz-Párraga, 2011). Scoring: Items are summed, with a total score from 11-44 and higher values represent a worse outcome (more pain interference in behavior).
Change from Baseline Numerical rating scale (NRS) at 6 and 12 weeks | Baseline (0 weeks), 6 weeks and 12 week
  The patient must rate his or her pain on a defined scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
Change from Baseline Boston Carpal Tunnel Questionnaire (BCTQ) at 6 and 12 weeks | Baseline (0 weeks), 6 weeks and 12 week
  The BCTQ measures self-reported functional status (BCTQ-F) and severity (BCTQ-S). The BCTQ-S consists of 11 questions, each question provides 5 response choices, from 1 (no symptoms) to 5 (most severe/often). The BCTQ-F includes 8 questions assessing difficulty with daily tasks. These responses are also scored on a 5-point scale (1-5).
Change from Baseline Hospital Anxiety and Depression Scale (HAD) at 6 and 12 weeks | Baseline (0 weeks), 6 weeks and 12 week
  Patient's emotional state will be evaluated by Hospital Anxiety and Depression Scale (HAD), which assess the level of anxiety and depression. Subscales and score range are Anxiety (0-21) and Depression (0-21). Scoring: items of each subscale are summed, indicating: 0-7 normality, 8-10 probably case, 11-21 anxiety or depression clinical case. Higher values represent a worse outcome.
Change from Baseline EQ-5D at 6 and 12 weeks | Baseline (0 weeks), 6 weeks and 12 week
  The EQ-5D is a self-assessed health-related quality of life questionnaire. The EQ-5D consists essentially of 2 pages: the EQ-5D description system and the visual analog scale (EQ VAS).
Hand diagrams | Baseline (0 weeks)
  To define total area marked for pain and numbness. The areas of the hand are marked by the patient and the marked area is quantified in square centimeters.
Change from Baseline Muscular endurance at 6 and 12 weeks | Baseline (0 weeks), 6 weeks and 12 week
  Maximum number of repetitions of rapid opening and closing of the hand until fatigue.
Patient Global Impression of Change Scale (PGICS) | 6 weeks
  The PGICS consists of two subscales, one categorical and one quantitative. The categorical scale is a 7-point verbal scale with the options "I have improved a lot" = 7, "I have improved a lot" = 6, "I have improved a little" = 5, "I am the same" = 4, "I have gotten a little worse" = 3, "I have gotten a lot worse" = 2, "I have gotten a lot worse" = 1.205-207 And, the quantitative scale consists of a line from 0 to 10, where 0 = much better and 10 = much worse.
Patient Global Impression of Change Scale (PGICS) | 12 weeks
  The PGICS consists of two subscales, one categorical and one quantitative. The categorical scale is a 7-point verbal scale with the options "I have improved a lot" = 7, "I have improved a lot" = 6, "I have improved a little" = 5, "I am the same" = 4, "I have gotten a little worse" = 3, "I have gotten a lot worse" = 2, "I have gotten a lot worse" = 1.205-207 And, the quantitative scale consists of a line from 0 to 10, where 0 = much better and 10 = much worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital la Florida, Santiago, Chile

REFERENCES:
- [Derived] Nunez-Cortes R, Cruz-Montecinos C, Torreblanca-Vargas S, Tapia C, Gutierrez-Jimenez M, Torres-Gangas P, Calatayud J, Perez-Alenda S. Effectiveness of adding pain neuroscience education to telerehabilitation in patients with carpal tunnel syndrome: A randomized controlled trial. Musculoskelet Sci Pract. 2023 Oct;67:102835. doi: 10.1016/j.msksp.2023.102835. Epub 2023 Jul 28. PMID 37572618